CLINICAL TRIAL: NCT06761443
Title: Based on a Randomized, Double-blind, Placebo-controlled Trial, we Evaluated the Safety and Efficacy of Pediococcus Acidilactici PA53 in Relieving Constipation in Adults
Brief Title: To Evaluate the Safety and Efficacy of Pediococcus Acidilactici PA53 in Relieving Constipation in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WK2024018
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Every day to Pediococcus acidilactici PA53 (30 billion CFU/day, 3g) intervention, for 8 weeks.
  Store in a cool and dry place.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Every day to give 3 g maltodextrin intervention for 8 weeks. Store in a cool and dry place.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study had last 8 weeks and each patient will make 3 visits (week 0, week 4, week 8).
  Arms: Probiotic
Dietary Supplement: Maltodextrin — The experimental phase of this study had last 8 weeks and each patient will make 3 visits (week 0, week 4, week 8).
  Arms: Placebo

SUMMARY:
To study the improvement of constipation symptoms, quality of life and mental state, intestinal function, intestinal hormones, inflammation and immunity, and intestinal flora of constipation subjects after 8-week intervention with Pediococcus acidilactici PA53.

ELIGIBILITY:
Inclusion Criteria:

1. Constipated subjects Subjects (less than 3 bowel movements per week and/or Bristol Scale Types 1 and 2); 2. Be able to complete the research according to the requirements of the test plan; 3. Subjects who have signed informed consent; 4. Subjects (including male subjects) have no family planning and voluntarily take effective contraceptive measures from 14 days before screening to 6 months after the end of the trial.

-

Exclusion Criteria:

1. Short-term use of items with similar functions to the subject, which affects the judge of the result;
2. Those who changed their diet type during the study period;
3. People with severe allergies and immune deficiencies;
4. Women who are pregnant, breastfeeding or planning to become pregnant;
5. Patients with serious diseases of cardiovascular, lung, liver, kidney and other vital organs, diabetes, thyroid disease, severe metabolic diseases, malignant tumors, and severe immune system diseases;
6. People who have used antibiotics in the past two weeks;
7. People with serious mental and mental illness;
8. Failure to eat the test sample as required, or failure to follow up on time, resulting in uncertain efficacy;
9. Other researchers judged it inappropriate to participate. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-05-25 (Estimated)

PRIMARY OUTCOMES:
Constipation symptom improvement | 8 weeks
  Assessing the improvement of constipation in patients using the Bristol Stool Form Scale (BSFS) . In this scale, higher scores indicate softer stool textures, closer to liquid consistency. Scores of 4, 5, and 6 are generally considered ideal stool characteristics.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China